CLINICAL TRIAL: NCT03135210
Title: The Impact of Lower Extremity Weight-Bearing Leg Exercise During the Pre-Ambulation Phase of Individuals Undergoing Extracorporeal Membrane Oxygenation
Brief Title: Leg Exercise During ECMO
Acronym: ECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1703M10081
Record Dates: First submitted 2017-04-21; First posted 2017-05-01 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Refractory Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: 24 total subjects will be recruited; 12 per group. Approximately 3-5 patients are admitted to UMMC each month who are undergoing ECMO and could be considered for study inclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Open-Chain Leg Exercise (Active Comparator): Individuals in the open-chain group will progress through standard mobility progression.
  Interventions: Other: Open-Chain Leg Exercise
- Closed-Chain Leg Exercise (Experimental): Individuals in the closed-chain group will progress through standard mobility exercises with the addition of closed-chain leg exercises using the MOVEO platform.
  Interventions: Device: Closed-Chain Leg Exercise

INTERVENTIONS:
Other: Open-Chain Leg Exercise — Individuals in the open-chain group will progress through standard mobility progression.
  Arms: Open-Chain Leg Exercise
Device: Closed-Chain Leg Exercise — Individuals in the closed-chain group will progress through standard mobility exercises with the addition of closed-chain leg exercises using the MOVEO platform.
  Other Names: Moveo Platform
  Arms: Closed-Chain Leg Exercise

SUMMARY:
Patients undergoing extracorporeal membrane oxygenation (ECMO) are at high risk for deconditioning and functional decline. The primary aim of this study is to assess the functional impact of leg exercise during the pre-ambulation phase in patients undergoing ECMO.

DETAILED DESCRIPTION:
The investigators are conducting this study to explore the impact of closed-chain leg exercise in individuals undergoing ECMO.

Aim 1: To determine if closed-chain leg exercise decreases the time to initial ambulation. The investgators hypothesize that adding leg exercise will decrease time to ambulation.

Aim 2: To determine the impact of closed chain leg exercise on functional ability. The investigators hypothesize that adding leg exercise will improve functional outcomes when added to an existing early mobilization program.

Aim 3: To determine the effect of closed chain leg exercise on hospital outcomes. The investigators hypothesize that hospital related outcomes will improve when leg exercise is added to an existing early mobilization program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory respiratory failure undergoing ECMO at the University of Minnesota Medical Center, Fairview.
* Able to follow 3 out of 3 one-step commands via protocol.
* Active Inpatient Physical Therapy Referral.
* ECMO delivery is veno-venous with internal jugular catheter.

Exclusion Criteria:

* Femoral catheter of any kind present
* Veno-arterial ECMO set-up
* Sedation such that self-consent is not attainable
* Medical instability, as determined by primary critical care physician

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda N LaLonde, DPT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-Chain Leg Exercise | Closed-Chain Leg Exercise
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-Chain Leg Exercise | Closed-Chain Leg Exercise | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 38 [27 to 49] | 52.5 [48 to 57] | 45.25 [27 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Ambulation
Description: Time to ambulation is measured as the number of days required for the participant to regain the ability to walk without the need for any kind of assistance. The unit of measure is days.
Time Frame: Baseline, to day 45 if applicable
Population: One participant in closed-chain leg exercise group expired after signing the consent form. Baseline data for this participant is included in the baseline characteristics section. Interventional data was not collected for this participant. All participants for whom outcome measure was collected are included in this analysis.
Measure: Mean (Full Range); unit: days
Arm/Group | Open-Chain Leg Exercise | Closed-Chain Leg Exercise
Number analyzed (Participants) | 2 | 1
days | 14.5 [11 to 18] | 15 [15 to 15]

ADVERSE EVENTS:
Time Frame: Participants are monitored for adverse events for the length of the study, up to 45 days following initiation of ECMO treatment.
Description: All participants were followed for adverse event collection.
Arm/Group | Open-Chain Leg Exercise | Closed-Chain Leg Exercise
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT03135210/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT03135210/ICF_001.pdf